CLINICAL TRIAL: NCT03538327
Title: Metabolic and Vascular Effects of Silybin in Hypertensive Patients With High One-hour Post-load Plasma Glucose: a Single Arm Pilot Study
Brief Title: Effects of Silybin in Hypertensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Maria Perticone, Principal Investigator, University Magna Graecia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UNICZ02
Record Dates: First submitted 2018-04-03; First posted 2018-05-29 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Hypertension
Keywords: essential hypertension; insulin resistance; silybin
MeSH Terms: conditions — Hypertension; Essential Hypertension; Insulin Resistance | interventions — Silybin

STUDY DESIGN:
Intervention Model Description: Pilot, single arm, interventional, longitudinal study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Silybin (Experimental): 50 Caucasian never-treated hypertensive outpatients, 27 males and 23 women, age range 42-60 years (mean+SD=52+7), showing normal glucose tolerance but 1-h post load plasma glucose >155 mg/dl, during the OGTT.
  Interventions: Drug: Silybin

INTERVENTIONS:
Drug: Silybin — After enrollment, all patients were encouraged to make lifestyle changes according with current guidelines, moreover it was also recommended to take silybin coniugated to vitamin E and phosphatidylcholine that shows higher intestinal absorption and bioavailability (Indena, IBI-Lorenzini spa Italy: Realsil®), as granules for oral solution at a dose of 3 g bid. Each subject was re-evaluated monthly performing a clinical examination to consider the opportunity of antihypertensive treatment. Finally, inflammatory, metabolic and hemodynamic parameters were assessed after 6 months of treatment. In particular, at the end of the follow-up period, a new OGTT was performed, to test the effects of silybin on glucose tolerance and IR status.

SUMMARY:
Background: Hypertensive patients with normal glucose tolerance (NGT) but 1-h post load plasma glucose >155 mg/dl (1-h high), during the oral glucose tolerance test (OGTT), show an unfavorable metabolic profile characterized by higher insulin resistance (IR), subclinical inflammation and multiple target organ damage. Experimental and clinical studies have demonstrated that silybin presents important anti-inflammatory and metabolic effects, improving IR and endothelial dysfunction. The present study aims to evaluate the effects of the complex silybin-vitamin E and phospholipids on inflammatory, metabolic and vascular parameters in NGT 1-h high hypertensive patients.

Methods: This is a pilot, single arm, interventional, longitudinal study in which the investigators have planned to enroll 50 Caucasian never-treated hypertensive outpatients, showing normal glucose tolerance but 1-h post load plasma glucose >155 mg/dl, during the OGTT.

DETAILED DESCRIPTION:
Insulin resistance (IR) represents a common pathophysiological mechanism of type 2 diabetes and arterial hypertension, both associated with the appearance and progression of cardiovascular disease (CVD).

Recently, it has been reported that a value of one-hour (1-h) post-load plasma glucose ≥155 mg/dL (1-h high), during an oral glucose tolerance test (OGTT), is able to identify subjects with normal glucose tolerance (NGT) but at high risk of incident type 2 diabetes; according with this, 1-h high NGT hypertensive patients show an unfavorable metabolic profile characterized by higher IR, subclinical inflammation and multiple target organ damage, similar to that observed in individuals with impaired glucose tolerance (IGT).

Experimental and clinical studies have demonstrated that silybin, the main active component extracted from the milk thistle, presents important anti-inflammatory, antifibrotic and metabolic effects, particularly, in the liver. In patients with non-alcoholic fatty liver disease (NAFLD), the complex silybin-vitamin E-phospholipids may improve all metabolic syndrome parameters, reducing IR and ameliorating glucose metabolism and liver histology. Given the common pathophysiological pathways shared by both cardiovascular and metabolic diseases, it's plausible that silybin may be protective also for tissues other than the liver, and in different clinical settings. According with this, silybin showed to markedly improve IR and endothelial dysfunction in an animal model of diabetes and obesity. On the basis of these considerations, the aim of this study was to evaluate the effects of the complex silybin-vitamin E and phospholipids (®Realsil) on inflammatory, metabolic and vascular parameters in a group of never treated 1-h high NGT hypertensive patients.

This is a pilot, single arm, interventional, longitudinal study for which the investigators have planned to enroll 50 Caucasian never-treated hypertensive outpatients, who resulted NGT with 1-h post load plasma glucose >155 mg/dl, during OGTT. All patients will undergo physical examination and review of their medical history. Causes of secondary hypertension will be excluded by appropriate clinical and biochemical tests. Other exclusion criteria are: history or clinical evidence of ischemic or valvular heart disease, congestive heart failure, peripheral vascular and chronic gastrointestinal diseases associated with malabsorption, chronic pancreatitis, history of any malignant or autoimmune disease, alcohol or drug abuse, liver or kidney failure, treatments able to modify glucose metabolism and smoking.

All subjects will undergo anthropometrical evaluation by measuring weight, height, body mass index (BMI) and waist. After 12-h fasting, a 75 g OGTT will be performed with 0, 30-, 60-, 90- and 120-min sampling for plasma glucose and insulin. Glucose tolerance status will be defined on the basis of OGTT using the World Health Organization (WHO) criteria.

Glucose, triglyceride, total and high density lipoprotein cholesterol (HDL-C) concentrations will be determined by enzymatic methods (Roche, Basel, Switzerland). Plasma insulin concentration will be determined with a chemiluminescence based assay (Immulite, Siemens, Italy). The minimum detectable concentration is 2 mIU/mL, and the maximal inter-assay coefficient of variation is 5.5%. Total serum insulin like growth factor (IGF)-1 concentrations will be measured by a chemiluminescent immunoassay (Nichols Institute Diagnostic, San Juan Capistrano, CA). The minimum detectable concentration is 0.03 mg/l, and the maximal inter-assay coefficient of variation is 7%. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels will be measured using the a-ketoglutarate reaction; and high sensitivity C reactive protein (hs-CRP) will be measured by automated instrument (CardioPhase_ hsCRP, Siemens, Italy). The intra-assay coefficient of variation for hs-CRP is <6%. Serum creatinine and uric acid (UA) will be measured in the routine laboratory by an automated technique based on the measurement of Jaffe chromogen and by the URICASE/POD (Boehringer Mannheim, Mannheim, Germany) method implemented in an autoanalyzer.

Insulin sensitivity The homeostasis model assessment (HOMA) index will be calculated as [fasting insulin (μU/mL) x fasting glucose (mmol/liter)]/22.5. Insulin sensitivity will be evaluated using the Matsuda index (insulin sensitivity index [ISI]), calculated as follows: 10,000/square root of [fasting glucose (mmol per liter) × fasting insulin (mU per liter)] × [mean glucose × mean insulin during OGTT]. The Matsuda index is strongly related to euglycemic-hyperinsulinemic clamp, which represents the gold standard test for measuring insulin sensitivity. The trapezoidal method will be used to calculate glucose and insulin area under curve (AUC) during the OGTT. Renal function will be evaluated by calculation of estimated-glomerular filtration rate (e-GFR), using the CKD-Epi equation.

Blood pressure measurements Readings of clinic blood pressure (BP) will be obtained in the left arm of the supine patients, after 5 min of quiet rest, with a mercury sphygmomanometer. Systolic BP (SBP) and diastolic BP (DBP) will be recorded at the first appearance (phase I) and the disappearance (phase V) of Korotkoff sounds. Baseline BP values will be the average of the last two of the three consecutive measurements obtained at intervals of 3 min, on three separate occasions at least 2 weeks apart. Patients with a clinic SBP>140 mmHg and/or DBP>90 mmHg will be defined as hypertensive, according with current guidelines. For the study protocol only patients with essential arterial hypertension of mild degree will be considered (SBP >140 mmHg and <160 mmHg and/or DBP >90 and <100 mmHg).

Arterial Stiffness and Central BP Measurements The evaluation of the arterial stiffness will be performed by the analysis of the shape and speed of the peripheral and central pressure wave. All studies will be performed in the supine position, in a quiet room with a constant temperature between 22°-24°C, after abstaining from cigarette smoking and food and alcohol intake in the 12 hours preceding the study. These measurements will be obtained by a validated system (SphygmocorTM; AtCor Medical, Sydney, Australia) that employs high-fidelity applanation tonometry (Millar) and appropriate computer software for the analysis of pressure wave (SphygmocorTM). Pressure calibration will be obtained through automatically, non-invasively recorded supine brachial artery BP of the dominant arm after a 30-minute rest (Dinamap Compact T; Johnson &Johnson Medical Ltd, Newport, UK). BP will be measured five times over 10 minutes and the mean of the last three measurements will be taken for calibration. Pressure wave recording will be performed at the radial artery of the dominant arm with the wrist softly hyperextended, and it is the average of single pressure waves recorded consecutively for eight seconds. Pressure wave recordings will be accepted only if variation of peak and bottom pressures of single pressure waves will be <5%. The central pressure wave will be automatically derived from the radial pressures by a built-ingeneralized transfer function. In addition, pressure wave measurement will be also obtained at the right carotid artery, as it is well known that central AI may be more accurately derived from this vascular site. Central waveforms will be further analysed to identify the time to peak/shoulder of the first (T1) and second (T2) pressure wave components during systole. The pressure at the peak/shoulder of T1 will be identified as outgoing pressure wave height (P1), the pressure at the peak/shoulder of T2 will be identified as the reflected pressure wave height (P2), either absolutely or as percent of ejection duration. Augmentation pressure (AP) will be defined as difference between P2-P1, and augmentation index (AI) as [AP/pulse pressure (PP)] * 100. Aortic pulse wave velocity (PWV) will be determined from carotid and femoral pressure waveforms. Carotid to femoral transit time (DT) will be computed from the foot-to-foot time difference between carotid and femoral waveforms. The distance between the surface markings of the sternal notch and femoral artery will be used to estimate the path length between the carotid and femoral arteries (L), and PWV computed as L/DT.

The protocol was approved by the local Ethical Committee (Comitato Etico Azienda Ospedaliera "Mater Domini") and informed written consent will be obtained from all participants. All the investigations will be performed in accordance with the principles of the Declaration of Helsinki.

Statistical analysis Continuous data are expressed as means + SD. For all variables, comparisons between baseline (T0) and post-treatment values (T6) will be performed using paired Student's t-test. The changes in all biomarkers in response to silybin intake will be expressed as mean and 95% CI, according with the CONSORT statement (21). Simple linear regression analysis will be performed to assess the relationship between variation in arterial stiffness indices (PWV, AI, AP), expressed as Δ of variation between baseline and follow-up (ΔT0-6) and the variation of metabolic and inflammatory covariates that significantly improved after the treatment (expressed as ΔT0-6). Thus, variables reaching statistical significance will be inserted in a stepwise multivariate linear regression model to assess the magnitude of their individual effect on Δ PWV, Δ AI and Δ AP, respecting the relationship of a variable every eight patients.

Differences will be assumed to be significant at P< 0.05. All comparisons will be performed using SPSS 20.0 statistical software for Windows (SPSS, Inc., Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive NGT patients with 1-h post load plasma glucose >155 mg/dl, during OGTT.

Exclusion Criteria:

* Secondary hypertension
* Ischemic or valvular heart disease
* Congestive heart failure
* Peripheral vascular disease
* Chronic gastrointestinal diseases associated with malabsorption
* Chronic pancreatitis
* History of any malignant or autoimmune disease
* Alcohol or drug abuse
* Liver or kidney failure
* Treatments able to modify glucose metabolism
* Smoking

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Improvement in fasting plasma glucose | six months after enrollment
  Fasting plasma glucose (mg/dL) will be measured after six months of treatment with silybin
Improvement in 2h post-load plasma glucose | Six months after enrollment
  2h post-load plasma glucose (mg/dL) will be determined after six months of treatment with silybin
Improvement in fasting insulin | Six months after enrollment
  Fasting insulin (mU/L) will be measured after six months of treatment with silybin
Improvement in total cholesterol | Six months after enrollment
  Total cholesterol (mg/dL) will be measured after six months of treatment with silybin
Improvement in HDL cholesterol | Six months after enrollment
  HDL-cholesterol (mg/dL) will be measured after six months of treatment with silybin
Improvement in LDL-cholesterol | Six months after enrollment
  LDL-cholesterol (mg/dL) will be measured after six months of treatment with silybin
Improvement in clinical SBP | six months after enrollment
  SBP (mmHg) will be measured after six months of treatment with silybin .
Improvement in clinical DBP (mmHg) | Six months after enrollment
  DBP (mmHg) will be measured after six months of treatment with silybin
Improvement in PP | Six months after enrollment
  PP will be measured after six months of treatment with silybin.
Improvement in PWV | Six months after enrollment
  PWV (m/s) will be measured after six months of treatment with silybin
Improvement in AI | Six months after enrollment
  AI will be measured after six months of treatment with silybin
Improvement in AP | Six months after enrollment
  AP (mmHg) will be measured after six months of treatment with silybin
Improvement in serum hs-CRP | Six months after enrollment
  Measurement of serum hs-CRPhs-CRP (mg/dL) will be measured after six moths of treatment with silybin

CONTACTS AND LOCATIONS:
Overall Officials: Maria Perticone, MD, Principal Investigator — Uniersity Magna Graecia of Catanzaro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loguercio C, Festi D. Silybin and the liver: from basic research to clinical practice. World J Gastroenterol. 2011 May 14;17(18):2288-301. doi: 10.3748/wjg.v17.i18.2288. PMID 21633595